CLINICAL TRIAL: NCT04954846
Title: Auswirkungen Eines Probiotischen Nahrungsergänzungsmittels Auf Das Darmmikrobiom Von Schlaganfallpatienten (PRISE)
Brief Title: A Randomized Double Blinded Placebo Controlled Study on the Effects of Dietary Supplementation With a Probiotic on Stroke Patients
Acronym: PRISE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Arthur Liesz, Professor Dr. med. Arthur Liesz, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRISE
Record Dates: First submitted 2021-06-18; First posted 2021-07-08 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Stroke, Ischemic; Dysbiosis
Keywords: Gut-Brain Axis; Probiotics; Food supplements; Microbiome
MeSH Terms: conditions — Ischemic Stroke; Dysbiosis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OMNi-BiOTiC SR-9 (Experimental): Treatment is taken twice a day for 3 months
  Interventions: Dietary Supplement: OMNi-BiOTiC SR-9
- Control (Placebo Comparator): Placebo is taken twice a day for 3 months
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: OMNi-BiOTiC SR-9 — The Probiotic contains the following ingredients:
  Maize Starch, Maltodextrin, Inulin, Potassium Chloride, Hydrolysed rice protein, Magnesium Sulphate, Fructooligosaccharides, Amylase, Manganese Sulphate
  Additionally, the following bacterial strains are included:
  Lactobacillus Casei W56, Lactobacillus Acidophilus W22, Lactobacillus Paracasei W20, Bifidobacterium lactis W51, Lactobacillus salivarius W24, Lactococcus lactis W19, Bifidobacterium lactis W52, Lactobacillus plantarum, Bifidobacterium bifidum W23
  Arms: OMNi-BiOTiC SR-9
Dietary Supplement: Placebo — The Placebo contains no bacterial strains, only the prebiotic ingredients found in OMNi-BiOTiC SR-9.
  Arms: Control

SUMMARY:
The aim of this study is to determine the effects of an intervention using a commercially available probiotic in a cohort of acute stroke patients. In order to determine this, a double blinded, randomised and placebo-controlled study design was chosen.

DETAILED DESCRIPTION:
Patients are recruited from the Stroke Unit of the Ludwig Maximilians University Munich within seven days of stroke onset. Recruited patients are then randomly assigned to either the Control or Treatment group and subsequently take the commercially available probiotic, or the placebo, twice a day for 3 months. At this point, study participants present themselves for routine clinical examination at the outpatient clinic of the Institute for Stroke and Dementia Research (ISD). During these examinations, blood and stool samples are collected for metabolomic and metagenomic analysis. Additionally, questionnaires concerning cognitive function (MOCA), depression (BDI) and general gastrointestinal status (GSRS-IBS) are completed.

Clinical data from both acute admission and three month follow-up are also collected for the purposes of this study.

Furthermore, members of the same household as the study participants are asked to donate a stool sample. These samples will be used to create a reference cohort for a paired matching approach with the Treatment and Control groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ischemic stroke with onset in past 7 days
* Treatment received in the Stroke Unit of the LMU University Hospital, location Großhadern

Exclusion Criteria:

* Chronic immunological disease
* Severe gastrointestinal disease
* Colectomy
* Artificial intestinal outlet (ostomy)
* Liver cirrhosis, pancreatitis, gastritis, cholecystitis (or other acute gastrointestinal diseases)
* Chronic alcohol abuse
* Terminal prognosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 157 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Alpha diversity, determined via Shannon index | 3 Months after stroke onset/Begin of diet supplementation
Alpha diversity, determined via phylogenetic diversity index | 3 Months after stroke onset/Begin of diet supplementation

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MOCA) | 3 Months after stroke onset/Begin of diet supplementation
  Range of achievable values is 0 - 31, low values are associated with impaired cognitive function
Becks Depression Inventory (BDI) | 3 Months after stroke onset/Begin of diet supplementation
  Range of achievable values is 0 - 63, high values are associated with mild (12-19), moderate (20-26) and severe (30-63) depression
National Institute of Health Stroke Scale (NIHSS) | 3 Months after stroke onset/Begin of diet supplementation
  Range of achievable values is 0 - 42, high values are associated with more advanced impairment due to stroke
Gastrointestinal Symptom Rating Scale for Irritable Bowel Syndrom (GSRS-IBS) | 3 Months after stroke onset/Begin of diet supplementation
  Range of achievable values is 13 - 91, high values are associated with more pronounced gastrointestinal symptoms (i.e. pain, diarrhea, discomfort)
Modified Rankin Scale (mRS) | 3 Months after stroke onset/Begin of diet supplementation
  Range of achievable values is 0 - 5, high values are associated with loss of mobility and autonomy
Beta diversity, determined via Bray-Curtis dissimilarity | 3 Months after stroke onset/Begin of diet supplementation
Beta diversity, determined via UniFrac | 3 Months after stroke onset/Begin of diet supplementation

CONTACTS AND LOCATIONS:
Locations (1):
- Ludwig Maximilian University Munich, University Hospital, Site Großhadern, Munich, Bavaria, Germany